CLINICAL TRIAL: NCT05383664
Title: Systemic Molecular Responses Caused by Exposure of Human Skin to Ultraviolet Light: a Pilot Study
Brief Title: Molecular Responses Caused by UV Exposure of Human Skin
Acronym: SMR-UV
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Access Business Group (Industry)
Collaborators: University of Michigan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Screening
Other Study IDs: CL22-04-EX01
Record Dates: First submitted 2022-05-09; First posted 2022-05-20 (Actual); Last update posted 2023-02-10 (Actual); Status verified 2023-02

CONDITIONS: Ultraviolet Light Burn
Keywords: Ultraviolet Light; Skin; Systemic Stress; Biomarkers

STUDY DESIGN:
Intervention Model Description: Sampling of blood biomarkers subsequent to successive bouts of UV-light exposure.
Masking Description: Baseline measurements serve as control; experimental design is sequential, no placebo or masking is necessary for the experimental design.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Clinical Screening (Experimental): Subjects will be screened for systemic blood markers responsive to 3-4 subsequent UV exposure over the course of 4-5 laboratory visits over the course of one week.
  Interventions: Other: Ultra Violet Light Exposure

INTERVENTIONS:
Other: Ultra Violet Light Exposure — Subjects will stand at the determined distance from the UV lamps facing towards them to achieve full body UV exposure. They will stand for the time indicated to achieve the appropriate dose. Each exposure will range from about 1 minute to 4.5 minutes to deliver a dose ranging from 0.22J/cm2 to 0.88J/cm2. Subjects will then rotate to irradiate their back side for the same time to achieve the same dose. On the second visit clinical examination will be conducted for erythema. If no erythema is apparent, the dosage on subsequent visits may increase to the max of 0.88 J/cm2.
  Other Names: UV Light Exposure

SUMMARY:
Pilot study to investigate the impact of exposure of human skin to low levels of UV light on blood markers related to stress in healthy women. Positive findings may serve to reframe the importance of skin health and skin care within the paradigm of holistic health and well-being.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is biologically female.
2. Subject age is 20-50 years, inclusive.
3. Subject has Fitzpatrick Skin Type I-III
4. Subject has a body mass index (BMI) of ≥ 18.5 and <30 kg/m2 at visit 1
5. Subject is willing to maintain habitual diet and physical activity patterns during the study period.
6. Subject does not smoke or use tobacco or nicotine-containing products of any kind, including vaping.
7. Subject has no health conditions that would prevent her from fulfilling the study requirements as judged by the study Investigator based on evaluation of medical history and routine laboratory test results.
8. Subject understands the study procedures and signs forms providing informed consent to participate in the study and authorization for release of relevant protected health information to the study Investigator.

Exclusion Criteria:

1. Subject is unwilling to avoid exposure to UVR, including natural sunlight, artificial UVR sources (e.g. tanning beds) for the duration of the study period.
2. Subject has a history of or is currently using any prescription medication, over-the-counter medication, natural product, dietary supplement, skin care product or cosmetic product that is known to produce abnormal responses to sunlight such as psoralens, hydrochlorothiazide, sulfa medications, certain antibiotics (tetracyclines, quinolones), amiodarone, furosemide, chlorpromazine.
3. Subject has a history of any abnormal responses to sunlight, such as a phototoxic or photoallergic response.
4. Subject has presence of any sunburn, suntan, scars, active dermal lesions, uneven skin tone, nevi, blemishes, moles, or other skin trait that, in the opinion of the Investigator, may interfere with study results.
5. Subject has a history or presence of a chronic skin condition or skin cancer.
6. Subject is biologically female who is pregnant, planning to be pregnant during the study period, or is lactating.
7. Subject has a recent history of use (within 4 weeks of visit 1) or is currently using any prescription and/or over-the-counter non-steroidal anti-inflammatory medication or immunosuppressive medications.
8. Subject has a recent history of use (within 4 weeks of visit 1) or is currently using any prescription and/or over-the-counter antihistamine known to increase sensitivity to sunlight or ultraviolet light.
9. Subject has used dietary supplements, other than a once-daily conventional multi-vitamin/multi-mineral supplement, within 4 weeks of visit 1 and is unwilling or unable to refrain from use for the duration of the study period.
10. Subject has history of use of omega-3-acid ethyl ester drug(s) or dietary supplement(s) containing fish oil, algal oil, krill oil, borage oil, DHA, or EPA within 4 weeks of visit 1 and is unwilling to discontinue use for the duration of the study period.
11. Subject has chronically consumed fatty fish (e.g., mackerel, salmon, trout, tuna, canned albacore tuna, sardines, haddock, cod, hake, halibut, sole, flounder, perch, black bass, swordfish, oysters, Alaskan king crab, shrimp, and/or lobster) in excess of 1 serving per week for 4 weeks of visit 1 and is unwilling to refrain from consumption throughout the study period.
12. Subject has chronically consumed foods rich in omega-3 fatty acids (e.g., flaxseed, chia seeds, walnuts, firm tofu, and/or fortified foods) within 4 weeks of visit 1 and/or is unwilling to discontinue use for the duration of the study period.
13. Subject has a history of use of antioxidant products, including foods, dietary supplements, and skin care products, within 4 weeks of visit 1 and is unwilling to discontinue use for the duration of the study period.
14. Subject has recent history of use (within 4 weeks of visit 1) or is a current user of herbal supplements, natural products, homeopathic remedies, and/or botanical supplements/extracts and is unwilling to discontinue use for the duration of the study period.
15. Subject has an active infection at visit 1 or use of antibiotics within 5 d of any clinic visit. For those with an active infection and/or using antibiotics, subjects must wait at least 5 d after the infection resolves or antibiotic use is complete to participate in a clinic visit.
16. Subject has a recent history (within 12 months of visit 1) or strong potential for alcohol or substance abuse. Alcohol abuse is defined as >14 drinks per week (1 drink = 12 oz beer, 5 oz wine, or 1½ oz distilled spirits).
17. Individual has a condition the study Investigator believes would interfere with her ability to provide informed consent or comply with the study protocol, which may confound the interpretation of the study results, or put the subject at undue risk.

Ages: 20 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2023-09-12 (Estimated); Study Completion 2024-09-12 (Estimated)

PRIMARY OUTCOMES:
Tumour Necrosis Factor alpha (ng/ml) | 1 week
  Biomarker of systemic stress
Interleukin 1 alpha (ng/ml) | 1 week
  Biomarker of systemic stress
Interleukin 6 (ng/ml) | 1 week
  Biomarker of systemic stress
Interleukin 10 (ng/ml) | 1 week
  Biomarker of systemic stress

SECONDARY OUTCOMES:
Dose frequency of UV light exposure | 1 week
  Level of UV light exposure to detect systemic response markers

OTHER OUTCOMES:
Adverse events | 1 week
  Safety and Tolerability
Heart rate | 1 week
  Safety and Tolerability
Blood pressure | 1 week
  Safety and Tolerability

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Leverett, Study Chair — Access Business Group; Gary Fisher, PhD, Principal Investigator — University of Michigan
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No
Data is collected will be used in development of protected and potentially patentable applications; therefore it is not planned to be made available to other researchers.